CLINICAL TRIAL: NCT04165408
Title: A Prospective, Non-Randomized, Single Arm Trial to Assess the Safety and Clinical Performance of the Contino®, a Urethral Insert, in Preventing Urinary Incontinence in Male Subjects With Sphincteric Incompetence
Brief Title: Trial to Assess the Safety and Clinical Performance of Contino® in Preventing Urinary Incontinence
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: One site still open but on hold due to financial issues. Enrollment will resume once payments are started up again. Other sites closed.
Sponsor: CMX Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMX-LF-2019-022
Record Dates: First submitted 2019-11-01; First posted 2019-11-18 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-08

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Device Use (Experimental): Only one arm
  Interventions: Device: Contino

INTERVENTIONS:
Device: Contino — The Contino® urethral insert is a self-administered licensed medical device, is inserted into the distal portion of the male urethra inhibiting the flow of urine. The Contino is self-inserted into the adult male urethra and is removed prior to urination. Much more than just a device, Contino® is an integrated solution that includes personalised fitting and support from incontinence specialists. It is made from highly specialised medical grade polymer, which has been extensively tested for biocompatibility.

SUMMARY:
This trial is to assess the safety and clinical performance of Contino device is preventing Urinary Incontinence in male subjects with Sphincteric Incompetence

DETAILED DESCRIPTION:
Sphincteric incompetence is most commonly found in men who have had radical prostatectomy (RP). RP is the most common treatment for localized high-risk Prostate Cancer in North America.

The Contino®, a urethral insert, was conceived by a prostate cancer survivor and worn for 10+ years without incident, and a First in Human clinical trial was completed without serious adverse event. The basis for this clinical trial is a post market clinical follow-up study. No drug treatment will be administered.

ELIGIBILITY:
Inclusion Criteria:

1. Male 18 years of age or older
2. Evidence of sphincteric incompetence as assessed by the Investigator
3. ECOG 0 or 1 performance status
4. Evidence of moderate to severe urinary incontinence as assessed by the Investigator, typically 2 or more protective garments or pads per day

Exclusion Criteria:

1. Inability to consistently insert the Contino® into his own urethra and remove it
2. Less than 2 months post radical prostatectomy for localized prostate cancer
3. History of significant incontinence that is other than stress incontinence
4. Evidence of neurogenic bladder dysfunction resulting in uncontrolled contractions
5. Untreated urethral stricture disease
6. Use of anticoagulant or antiplatelet medications excluding low-dose ASA (in the opinion of the Investigator)
7. Any cardiac condition that requires the use of pre-procedure antibiotic prophylaxis such as a mechanical valve (in the opinion of the Investigator)
8. Body Mass Index (BMI) greater than 32 kg/m2 (in the opinion of the Investigator provided the subject is able to insert & remove the device)
9. Known immune deficiency either due to disease or medications (in the opinion of the Investigator)
10. Uncontrolled diabetes (in the opinion of the Investigator)
11. An UTI (in the opinion of the Investigator)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 25 (Estimated)
Dates: Start 2019-11-19 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
To establish the safety of the Contino® | 14 Months
  safety is characterized by the absence of complications
To establish the clinical performance of the Contino® | 14 Months
  Clinical performance is characterized by the ability to stop involuntary urine flow
Change from baseline in the ICIQ-SF score | 14 Months
  At Visit Days 30 and 60
Change from baseline in the weight of the protective pads | 14 Months
  At Visit Days 30 and 60

SECONDARY OUTCOMES:
Level of ease of use inserting the Contino® from the Follow-up Questionnaire | 14 Months
  Level of comfort measurement
Level of ease of use removing the Contino® from the Follow-up Questionnaire | 14 Months
  Level of comfort measurement
Number of subjects with newly observed urinary function improvements | 14 Months
  including (but not limited to): being able to urinate independently for the first time since prostate surgery, return of urge to void and sensation of full bladder, better urinary stream, reduced time urinating from the follow up questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Dean Elterman, MD, Principal Investigator — University Urology Associates
Locations (2):
- Canada (2):
  - The Fe/Male Health Centres, Oakville, Ontario
  - Dr. Dean Elterman, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No